CLINICAL TRIAL: NCT03938168
Title: PAIN PAD Histological and Molecular Mechanisms of Pain in Patient With Chronic Pain From Adhesions
Brief Title: Histological and Molecular Mechanisms of Pain in Patient With Chronic Pain From Adhesions
Acronym: PAIN PAD
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Maastricht University Medical Center (Other); Maas Hospital Pantein (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-4801
Record Dates: First submitted 2019-05-01; First posted 2019-05-06 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Tissue Adhesion; Chronic Pain; Surgery
MeSH Terms: conditions — Tissue Adhesions; Chronic Pain | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples from adhesions are taken. Fecal samples are taken for microbioma analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pain patients: 30 patients eligible for adhesiolysis because of chronic adhesion-related pain. Patients are recruited at the RadboudUMC, MUMC+ and Pantein hospital departments of surgery. These are patients with chronic pain after previous abdominal surgery who have been selected for operative treatment after evaluated with CineMRI. CineMRI is used to map adhesions. This technique has been established to provide insight in localization of adhesions in relation to the pain, and risk of bowel injury based on extensiveness of adhesions.
  Interventions: Diagnostic Test: Biopsy, fecal sample
- Control group: The control group will comprise of 30 patients undergoing an abdominal reoperation during which adhesiolysis has to be performed for reasons other than chronic adhesion-related pain.
  Interventions: Diagnostic Test: Biopsy, fecal sample

INTERVENTIONS:
Diagnostic Test: Biopsy, fecal sample — Preoperatively and at 12 months after surgery, patients will obtain a fecal stool sample for microbioma analysis. Adhesions that are cut and released to acquire access to the operative field are stored for molecular and histological analyses.

SUMMARY:
11-20% of patients undergoing abdominal surgery develop chronic abdominal pain. Adhesions are a common cause of chronic pain following surgery. Adhesions develop after up to 90% of laparotomies and 70% of laparoscopic surgeries. Obviously, not all adhesions cause pain. It is still poorly understood why adhesions cause pain in some patients, while other patients with adhesions experience no pain.

In this study we explore possible mechanism through which adhesions might cause pain. For this purpose we will assess expression of molecular mediators (such as TRPV-1, SP, and the neurokinin receptor), histological characteristics, and fecal microbioma that might be associated with pain.Expression of these factor will be compared to sample from 30 patients with chronic pain attributed to adhesions, and 30 patients undergoing a reoperation with adhsiolysis for reasons unrelated to pain.

DETAILED DESCRIPTION:
Introduction and rationale:

11-20% of patients undergoing abdominal surgery develop chronic abdominal pain. Adhesions are the most common cause of chronic abdominal complaints after surgery. Chronic pain from adhesions has devastating consequences for quality of life, and one in three patients with pain from adhesions is opioid dependent.

Adhesions develop after up to 90% of laparotomies and 70% of laparoscopic surgeries. Obviously, not all adhesions cause pain. It is still poorly understood why adhesions cause pain in some patients, while other patients with adhesions experience no pain.

In a recent study we demonstrated that in selected patients adhesion-related pain can effectively be treated by operation with adhesiolysis and application of an adhesion barrier. However, almost 50% part of patients with adhesion-related pain are not considered a candidate for surgical treatment, for various reasons.

Exploring the mechanisms that contribute to development of pain in patients with adhesions could provide novel targets for medical therapies. These could greatly benefit many patients suffering from adhesion- related pain. Two factors that might explain why some patients with adhesions develop chronic pain are activation of molecular mechanisms involved in chronic pain and stimulation of nerve fibers present in adhesions. Specifically type C nerve fibres are associated with development of neuropathic pain. Further we will also explore differences in microbioma, which has recently been demonstrated to have an important role in a variety of abdominal conditions.

Adhesion formation at the molecular level involves a complex interaction of mediators. One such mediator that might link adhesion formation to nociception is the pro-inflammatory peptide substance P.(1) Substance P in turn is mediated by Transient Receptor Potential Vanilloid (TRPV1), which is known to be upregulated in many conditions associated with chronic pain. There is currently much research in developing new analgesics targeting this receptor. Previous studies have shown that nerve fibres can be present in adhesive tissue. Presence of such fibres, and especially type C fibres might be responsible for a neuropathic type of pain. Stimulation of TRPV1 might also activate type C nerve fibre endings.

Objective:

Quantify and compare expression of molecular mediators (such as TRPV-1, SP, and the neurokinin receptor) and histological characteristics of adhesions from patients with postoperative adhesions with and without chronic abdominal pain. Comparison of microbioma in fecal samples between patients with adhesions with and without chronic abdominal pain

Study design:

This is a prospective observational cohort study.

Study population:

30 patients eligible for adhesiolysis because of chronic adhesion-related pain. Patients are recruited at the RadboudUMC, MUMC+ and Pantein hospital departments of surgery. These are patients with chronic pain after previous abdominal surgery who have been selected for operative treatment after evaluated with CineMRI. CineMRI is used to map adhesions. This technique has been established to provide insight in localization of adhesions in relation to the pain, and risk of bowel injury based on extensiveness of adhesions. The control group will comprise of 30 patients undergoing an abdominal reoperation during which adhesiolysis has to be performed for reasons other than chronic adhesion-related pain.

Study procedures:

Prior to surgery patients are requested to take a stool sample. During surgery histological samples of adhesions will be taken during adhesiolysis in both groups. In the control group histological samples of adhesions will only be taken if it does not require extension of the incision and if it is not accompanied with additional risk of intraoperative complications other than necessary for their planned surgery.

Main study parameters/endpoints:

Primary outcome mRNA expression levels of TRPV1 by quantitative polymerase chain reaction (qPCR) compared between patients with and without chronic pain. Secondary outcomes are TRPV1 protein levels (measured by Westernblot), SP, and neurokinin expression, and the amount and types of nerve fibres found at histological assessment. Further we will explore microbioma in feca samples.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Taking fecal and histological samples for this study does not result in additional operative risk. Adhesiolysis is often performed during any type of abdominal reoperation. Histological samples in controls are only taken from adhesions that are easily accessible and not from dense adhesions in close proximity to bowel or other vulnerable organs. No additional adhesiolysis apart from biopsy will be performed.

ELIGIBILITY:
In order to be eligible to participate patients with chronic pain, must meet all of the following criteria:

* Abdominal pain for more than 12 months after last surgery
* Insufficient improvement of pain after conservative treatments for at least 6 months
* Pre-operative work-up with cineMRI showing expected beneficial outcomes of adhesiolysis, in accordance to our current standard practice for adhesion-related pain.

Inclusion criteria for controls:

* Patients between 18 and 75 years old scheduled for elective abdominal reoperation
* No present chronic abdominal pain
* No other diseases or syndromes that cause chronic pain (e.g. rheumatic arthritis)

Exclusion criteria

A potential subject with chronic pain will be excluded from participation in this study in the following cases:

* Contra-indications for general anaesthesia and re-operation
* Inability to acquire informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic abdominal pain after surgery is a frequent condition.(13) At present the RadboudUMC, MUMC+, and Pantein hospital departments of surgery annually evaluate 60-80 patients each for chronic pain by cineMRI. Between 30-40 of these patients are expected to undergo surgical treatment. Yearly between 600-700 patients will undergo an elective abdominal reoperation at the participating departments of surgery. Thus there is ample surgical volume for this study.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
TRPV-1 | during surgery
  mRNA expression levels of TRPV1 by quantitative polymerase chain reaction (qPCR)

SECONDARY OUTCOMES:
TRPV-1 protein | during surgery
  TRPV1 protein levels (measured by Westernblot)
SP | during surgery
  mRNA expression levels of Substance P
NK-1 | during surgery
  mRNA expression levels of Neurokinin 1
Nerve fibers | during surgery
  Histological assessment for the presence of nerve fibers
Microbioma | 12 months
  alpha and beta diversity of Fecal microbioma pre-operative and at 12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Richard P ten Broek, MD, PhD, Principal Investigator — Radboud University Medical Center; Harry van Goor, MD, PhD, Study Director — Radboud University Medical Center; Richard P ten Broek, MD, PhD, Study Chair — Radboud University Medical Center
Locations (3):
- Netherlands (3):
  - Maasziekenhuis Pantein, Boxmeer, Gelderland
  - Radboud University Medical Center, Nijmegen, Gelderland
  - Maastricht Universitair Medisch Centrum+, Maastricht, Limburg

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared upon reasonable request through DANS easy archive
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 12 months after publication of primary results

REFERENCES:
- [Background] van den Beukel BAW, Stommel MWJ, van Leuven S, Strik C, IJsseldijk MA, Joosten F, van Goor H, Ten Broek RPG. A Shared Decision Approach to Chronic Abdominal Pain Based on Cine-MRI: A Prospective Cohort Study. Am J Gastroenterol. 2018 Aug;113(8):1229-1237. doi: 10.1038/s41395-018-0158-9. Epub 2018 Jun 27. PMID 29946174
- [Background] Reed KL, Fruin AB, Bishop-Bartolomei KK, Gower AC, Nicolaou M, Stucchi AF, Leeman SE, Becker JM. Neurokinin-1 receptor and substance P messenger RNA levels increase during intraabdominal adhesion formation. J Surg Res. 2002 Nov;108(1):165-72. doi: 10.1006/jsre.2002.6533. PMID 12443729
- [Background] ten Broek RP, Issa Y, van Santbrink EJ, Bouvy ND, Kruitwagen RF, Jeekel J, Bakkum EA, Rovers MM, van Goor H. Burden of adhesions in abdominal and pelvic surgery: systematic review and met-analysis. BMJ. 2013 Oct 3;347:f5588. doi: 10.1136/bmj.f5588. PMID 24092941
- [Background] Keszthelyi D, Troost FJ, Jonkers DM, Helyes Z, Hamer HM, Ludidi S, Vanhoutvin S, Venema K, Dekker J, Szolcsanyi J, Masclee AA. Alterations in mucosal neuropeptides in patients with irritable bowel syndrome and ulcerative colitis in remission: a role in pain symptom generation? Eur J Pain. 2013 Oct;17(9):1299-306. doi: 10.1002/j.1532-2149.2013.00309.x. Epub 2013 Mar 25. PMID 23529955
- [Background] Scotland RS, Chauhan S, Davis C, De Felipe C, Hunt S, Kabir J, Kotsonis P, Oh U, Ahluwalia A. Vanilloid receptor TRPV1, sensory C-fibers, and vascular autoregulation: a novel mechanism involved in myogenic constriction. Circ Res. 2004 Nov 12;95(10):1027-34. doi: 10.1161/01.RES.0000148633.93110.24. Epub 2004 Oct 21. PMID 15499026